CLINICAL TRIAL: NCT00753935
Title: Evaluation of Aspirin Resistance at a Molecular Level in Aspirin-Treated Patients With Coronary Artery Disease
Brief Title: Aspirin Resistance in Coronary Artery Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 040065; 5P50HL081009-03 (NIH)
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: aspirin; aspirin resistance; aspirin nonresponse; cyclooxygenase; thromboxane; oxidative stress
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enteric-coated aspirin (Experimental): patients received enteric-coated aspirin 81 mg qd for 2 weeks
  Interventions: Drug: enteric-coated aspirin
- Chewable aspirin (Active Comparator): Patients received chewable aspirin 81 mg qd for 2 weeks
  Interventions: Drug: Chewable aspirin

INTERVENTIONS:
Drug: enteric-coated aspirin — enteric-coated aspirin 81mg daily for 2 weeks
  Other Names: acetylsalicylic acid
  Arms: Enteric-coated aspirin
Drug: Chewable aspirin — chewable aspirin 81mg daily for 2 weeks
  Other Names: acetylsalicylic acid
  Arms: Chewable aspirin

SUMMARY:
The purpose of this study is to evaluate possible mechanisms of aspirin resistance at a molecular level in aspirin-treated patients with coronary artery disease. We hypothesize that certain patient characteristics associate with aspirin resistance. In addition, we will compare the effects of enteric-coated aspirin and chewable aspirin.

DETAILED DESCRIPTION:
Aspirin is commonly used for its antithrombotic effects in patients at risk for cardiovascular events. Its primary mechanism of action is the irreversible acetylation of platelet cyclooxygenase-1, thereby inhibiting platelet production of thromboxane A2, a potent vasoconstrictor and activator of platelets. Thromboxane A2, the major product of cyclooxygenase cytochrome oxidase (COX-1) in platelets, induces platelet aggregation. Thromboxane B2 is an inactive metabolite/product of thromboxane A2. This primary outcome measures the extent of inhibition of platelet COX-1 by measuring the amount of the metabolite thromboxane B2 in serum.

Previous studies have demonstrated that many patients have recurrent events despite treatment with aspirin, which has been termed "aspirin resistance" or "aspirin nonresponse." This study addresses some of the possible mechanisms for aspirin nonresponse; specifically, we will test the hypothesis that aspirin nonresponse results from states that produce high peroxide concentrations ("oxidative stress") in platelets. In addition, we will evaluate the effect of enteric coating on the pharmacologic efficacy of aspirin in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* On aspirin 81-325mg daily at time of enrollment
* Documented stable coronary artery disease or > 6 months after coronary artery bypass grafting or interventional cardiac procedure
* Written informed consent

Exclusion Criteria:

* Pre-menopausal female
* Renal disease (creatinine >= 2 mg/dl)
* Anemia (Hematocrit < 30%)
* Thrombocytopenia (platelet count < 135,000/ul)
* Use of NSAIDs or coxibs within the previous 2 weeks
* Concurrent use of other anti-platelet agents
* Uncontrolled hypertension (systolic BP > 180 mmHg)
* Decompensated congestive heart failure
* Recent coronary syndrome (< 6 months)
* History of significant GI bleeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2006-06; Primary Completion 2011-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Taylor, MD, MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Result] Smith JP, Haddad EV, Taylor MB, Oram D, Blakemore D, Chen Q, Boutaud O, Oates JA. Suboptimal inhibition of platelet cyclooxygenase-1 by aspirin in metabolic syndrome. Hypertension. 2012 Mar;59(3):719-25. doi: 10.1161/HYPERTENSIONAHA.111.181404. Epub 2012 Feb 6. PMID 22311905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enteric-coated Aspirin | Chewable Aspirin
Started | 45 | 47
Completed | 45 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enteric-coated Aspirin: patients with coronary artery disease received enteric-coated aspirin 81 mg qd for 2 weeks
- Chewable Aspirin: Patients with coronary artery disease received chewable aspirin 81 mg qd for 2 weeks
- Total: Total of all reporting groups
Arm/Group | Enteric-coated Aspirin | Chewable Aspirin | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Continuous [Mean (Full Range); unit: years] | 62 [56 to 69] | 68 [59 to 75] | 65 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 33 | 33 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 36 | 42 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 45 | 47 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Thromboxane B2
Description: Thromboxane A2, the major product of cyclooxygenase cytochrome oxidase (COX-1) in platelets, induces platelet aggregation. Thromboxane B2 is an inactive metabolite/product of thromboxane A2. This primary outcome measures the extent of inhibition of platelet COX-1 by measuring the amount of the metabolite thromboxane B2 in serum.
Time Frame: after 2 weeks on aspirin
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Enteric-coated Aspirin | Chewable Aspirin
Number analyzed (Participants) | 45 | 47
ng/mL | 5.02 [3.36 to 7.86] | 2.78 [1.60 to 4.76]
Statistical Analysis 1: Comparison: Enteric-coated Aspirin vs Chewable Aspirin; Test type: Superiority; p = 0.005, Wilcoxon rank-sum

ADVERSE EVENTS:
Time Frame: 2 years and 11 months
Arm/Group | Enteric-coated Aspirin | Chewable Aspirin
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47
Other Adverse Events (participants affected / at risk) | 0/45 | 0/47

LIMITATIONS AND CAVEATS:
There are no limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No